CLINICAL TRIAL: NCT05811975
Title: IIT Clinical Trial on Tolerance, Safety, and Preliminary Efficacy of KSX01-TCRT Injection in Solid Tumor Subjects
Brief Title: KSX01-TCRT Injection Project in Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: TCRx Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSX01-M101
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: TCR-T Cells; Refractory Solid Tumors; Relapsed Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental): Drug: KSX01 injection individualization TCR-T cell injection
  Interventions: Drug: KSX01-TCRT injection

INTERVENTIONS:
Drug: KSX01-TCRT injection — individualization TCR-T cell injection

SUMMARY:
1) Safety and efficacy of TCR-T cells in subjects with refractory/relapsed solid tumors. 2) The activation and proliferation of TCR-T cells in the subject, and the survival time.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary participation in clinical research; Fully understand the study and voluntarily sign an informed consent form; Willing to follow and capable of completing all test procedures.
* 2) Age: 18 to 70 years old (including boundary value).
* 3) Malignant solid tumors that have failed standard treatment or currently have no standard treatment available.
* 4) Patients with tumor lesions that can be punctured and can be screened for a pharmaceutically acceptable TCR sequence can be enrolled in the study.
* 5) Remission from previous surgical or treatment related adverse events to a level of 0-1, stable, or acceptable for inclusion/exclusion criteria (according to NCI CTCAE Version 5.0), or to an acceptable level for inclusion/exclusion criteria; Except for other toxicity that researchers believe does not pose a safety risk to the subject, such as hair loss, pigmentation, and peripheral neuropathy.
* 6) Adequate organ function (without medical support such as blood transfusion, granulocyte colony stimulating factor, etc. during pre harvest and baseline periods) is defined as follows:
* 6.1) Blood system:
* 6.1.1) Hemoglobin 90 g/L (no blood transfusion or erythropoietin treatment within 14 days before the first administration);
* 6.1.2) The absolute value of neutrophils is 1.5 109/L (no treatment with granulocyte colony stimulating factor or granulocyte macrophage colony stimulating factor within at least 14 days before chemotherapy);
* 6.1.3) Platelet count is 100 109/L in the absence of significant liver lesions (primary or metastatic), or 75 109/L in the presence of liver lesions (no platelet transfusion, thrombopoietin, or interleukin-11 treatment was received within 14 days before the first administration);
* 6.1.4) Absolute lymphocyte count (ALC) 0.7 109/L;
* 6.2) Liver function:
* 6.2.1) Total bilirubin (TBIL) ≤ 2.0 in the absence of significant liver lesions (primary or metastatic) × Upper limit of normal (ULN), subjects with liver lesions or Gilbert disease ≤ 3 × ULN；
* 6.2.2) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 × ULN (liver metastasis or hepatocellular carcinoma can be ≤ 5 × ULN）； Alkaline phosphatase (ALP) ≤ 2.5 × ULN (bone metastasis subject, ALP ≤ 5 × ULN）；
* 6.3) Renal function:
* 6.3.1) Creatinine clearance ≥ 50 ml/min (Cockcroft Gault formula: ([140 age] × Body weight [kg] × [0.85, female only])/(72 × Creatinine (mg/dl));
* 6.3.2) Qualitative determination of urinary protein ≤ 1+; If the qualitative analysis of urine protein is ≥ 2+, a 24-hour urine protein quantitative test is required. If the 24-hour urine protein quantitative analysis is<1 g, it is acceptable;
* 6.4) Coagulation function: Activated partial thromboplastin time and international standardized ratio of 1.5 in patients who did not receive anticoagulant therapy × ULN, or patients receiving anticoagulation therapy, have a stable anticoagulation treatment regimen; Patients with liver metastasis or liver cancer are acceptable 2 × ULN。
* 7) The Eastern United States Cancer Collaborative Group (ECOG) score for physical fitness is 0-1.
* 8) The expected survival period is ≥ 12 weeks.
* 9) According to the RECIST 1.1 standard, there is at least one evaluable lesion (dose increasing stage) or measurable lesion (dose expanding stage).
* 10) After evaluation, sufficient PBMC cells can be collected from the subjects to prepare autologous TCR-T cells; The peripheral superficial venous blood path of the subject is unobstructed, suitable for single blood collection and separation, with sufficient venous access to collect cells, and can meet the requirements of intravenous infusion.
* 11) After evaluation, the prepared autologous TCR-T cells are sufficient in quantity and qualified in quality, and can be used for corresponding doses of clinical reinfusion.
* 12) "The blood pregnancy test for women of childbearing age within 7 days before the first cell transfusion was negative, and the subjects of childbearing age used medically approved contraceptives from the beginning of research treatment (chemotherapy) until 1 year after the last cell transfusion, and no eggs were recovered during this period.".
* 13) Male subjects are willing to take medically approved contraceptive measures within 6 months after signing the informed consent form and the last cell transfusion, and do not donate sperm during this period.

Exclusion Criteria:

* 1) A history of severe allergic diseases, allergies to severe drugs (including unlisted investigational drugs), or known allergies to any component of the drugs recommended for use in this protocol (including pre-treatment drugs).
* 2) Persons who have previously received treatment with other cell/gene products.
* 3) Evidence of significant bleeding or coagulation disorders or other significant bleeding risks:
* 3.1) Previous history of intracranial hemorrhage or spinal cord hemorrhage;
* 3.2) Tumor lesions that invade large blood vessels and have a significant risk of bleeding;
* 3.3) Thrombosis or embolism occurred within 6 months before cell transfusion;
* 3.4) Clinically significant hemoptysis or tumor bleeding occurred within 1 month before cell reinfusion;
* 3.5) Within 2 weeks before cell reinfusion, anticoagulation therapy for therapeutic purposes has been used (except for those requiring a stable treatment regimen and judged appropriate by the researcher).
* 4) Within 28 days before enrollment, there were no healed wounds, ulcers, or fractures.
* 5) The following treatments or drugs have been received before enrollment, pre harvest, pre clearance, or cell reinfusion:
* 5.1) Have received any live or attenuated vaccine within 4 weeks before enrollment, or are expected to receive live or attenuated vaccine during the study period;
* 5.2) Preharvest use of any cytotoxic chemotherapy or small molecule targeted therapy<2 weeks or 5 half lives, whichever is longer;
* 5.3) Have undergone major surgery (excluding diagnostic surgery) within 4 weeks before single collection, or are expected to undergo major surgery during the study period;
* 5.4) Planned systemic use (if long-term use is expected) of systemic steroids (>10 mg/day of prednisone or equivalent), hydroxyurea, and immunomodulators (e.g.: α or γ Interferons, GM-CSF, mTOR inhibitors, cyclosporin, thymosin, etc.), this standard is not applicable when the following conditions occur:

  * Intranasal, inhalation, topical steroids, or local steroid injections (such as intra articular injections);
  * Physiological doses of systemic steroids as an alternative therapy (such as physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction);
  * Steroids are used as prophylaxis for hypersensitivity reactions (such as computed tomography (CT) prophylaxis).
* 5.5) The washout period of previous anticancer treatment before the first administration of the study drug is insufficient, as defined below:

  * Any cytotoxic chemotherapy or small-molecule targeted therapy<2 weeks or 5 half lives, whichever is shorter, except for clearance chemotherapy;
  * Endocrine therapy<3 weeks;
  * Monoclonal antibody or other biological therapy<3 weeks;
  * Herbal therapy with anti-tumor indications<2 weeks;
  * Whole brain radiotherapy<2 weeks, or stereotactic brain radiotherapy<1 week;
  * More than 30% of bone marrow radiotherapy or accompanied by wide field irradiation for<4 weeks, or palliative radiotherapy for<2 weeks.
* 6) Patients with systemic bone metastases.
* 7) A history of leptomeningeal cancer.
* 8) Brain metastases or spinal cord compression, unless asymptomatic, or symptoms stabilize after treatment and do not require treatment with steroids and anticonvulsants for at least 2 weeks prior to the first administration of the study drug.
* 9) Presence of any form of primary immune deficiency.
* 10) Subjects with any active autoimmune disease, or a history of autoimmune disease, and expected recurrence (including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease (such as Crohn's disease, ulcerative colitis), vasculitis, invasive lung disease, and asthma requiring medical intervention with bronchodilators). The following cases are excluded: type 1 diabetes; Skin diseases that do not require systemic treatment [such as vitiligo, psoriasis, alopecia, Grave's disease, Hashimoto's disease, psoriasis patients]; Hypothyroidism requiring only hormone replacement therapy; Asthma that has completely remitted in childhood does not require any intervention in adulthood; Or other people who are not expected to have a relapse without external triggers.
* 11) Active liver or biliary disease (excluding Gilbert syndrome or asymptomatic gallstones, liver metastases, or other stable chronic liver disease, as assessed by the investigator).
* 12) Within 6 months before cell reinfusion, the following conditions occurred: myocardial infarction, severe/unstable angina, clinically significant arrhythmias requiring clinical intervention, cerebrovascular accident/stroke, transient ischemic attack, subarachnoid hemorrhage, and cardiac insufficiency with a New York Heart Association (NYHA) rating of ≥ II.
* 13) There is currently uncontrolled pleural, pericardial, and abdominal effusion.
* 14) Before cell reinfusion, there are:
* 14.1) Congenital long QT syndrome;
* 14.2) Using a cardiac pacemaker;
* 14.3) Received coronary artery reconstruction;
* 14.4) Acute coronary syndrome (angina pectoris or myocardial infarction, within 6 months before signing the informed consent form);
* 14.5) The electrocardiogram showed clinically significant abnormalities or an average QTcF of>450 ms for men and>470 ms for women (>480 ms for patients with bundle branch block (BBB)) in three consecutive times (at least 5 minutes between each time interval);
* 14.6) Severely uncontrollable diabetes;
* 14.7) Hypertension with poor drug control (systolic blood pressure>160 mmHg and/or diastolic blood pressure>90 mmHg);
* 14.8) Severe aortic stenosis or symptomatic mitral stenosis;
* 14.9) Interstitial pneumonia or pulmonary fibrosis can be seen on chest radiographs (subjects with pneumonia due to radiation are not excluded, but they cannot rely on oxygen);
* 14.10) Any other disease that the researcher believes will impair the subject's tolerance to the treatment regimen or significantly increase the risk of complications;
* 15) During screening or before cell transfusion, fever of unknown origin>38.5 ° C occurred (according to the judgment of the researcher, fever caused by tumor can be included in the group).
* 16) There are severe active viral and bacterial infections, or uncontrolled systemic fungal infections within 4 weeks prior to enrollment, single collection, and pre treatment with cleaning and administration.
* 17) Virological examination results (HIV, Treponema pallidum antibody Tp-Ab) were positive.
* 18) Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive, and hepatitis B virus DNA (HBV-DNA) is higher than the lower limit of detection in the research center; HCV-Ab is positive and HCV-RNA is higher than the lower detection limit of the research center.
* 19) It is expected that any other form of anti-tumor drug treatment will be required during the study period after cell transfusion.
* 20) There is a known history of organ transplantation.
* 21) Women during pregnancy or lactation.
* 22) Known history of alcohol abuse, psychotropic substance abuse, or drug abuse.
* 23) Have a clear history of neurological or mental disorders, such as epilepsy, dementia, schizophrenia, etc.
* 24)According to the judgment of the researcher, the underlying condition of the subject may increase the risk of receiving treatment with the investigational drug, or may cause confusion in the interpretation of the toxic reactions and adverse events that occur.
* 25) Other situations where the researcher considers it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Subject safety | about 2 years
  Number of participants with treatment-related adverse events assessed by CTCAE v4.0.
tumor efficacy | about 2 years
  Changes in overall tumor diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ma, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The first affiliated hospital of Guang Xi medical university, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No